CLINICAL TRIAL: NCT00625170
Title: Metabolic Effects of Subchronic Dopamine D2 Receptor Blockade by Antipsychotic Drugs in Healthy Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Dutch Diabetes Research Foundation (Other)
Responsible Party: Prof. Hanno Pijl, LUMC
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: P03.136
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Last update posted 2008-02-28 (Estimated); Status verified 2004-03

CONDITIONS: Insulin Resistance; Dyslipidemia
Keywords: Antipsychotics; Olanzapine; Haloperidol; Insulin resistance; Dyslipidemia
MeSH Terms: conditions — Insulin Resistance; Dyslipidemias | interventions — Olanzapine; Haloperidol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Healthy men
  Interventions: Drug: olanzapine
- 2 (Active Comparator): Healthy men with a positive family anamneses of schizophrenia
  Interventions: Drug: olanzapine; Drug: Haloperidol

INTERVENTIONS:
Drug: olanzapine — olanzapine 10 mg/day for 8 days
  Other Names: Zyprexa
Drug: Haloperidol — haloperidol 3 mg/day for 8 days
  Arms: 2

SUMMARY:
We hypothesized that short-term treatment with AP drugs induces insulin resistance through a mechanistic route that is independent of weight gain and that atypical drugs exert stronger effects than typical compounds in this respect. We therefore treated healthy non-obese men with olanzapine (atypical AP) or haloperidol (typical AP) for 8 days, and studied the impact of these interventions on glucose and lipid metabolism by hyperinsulinemic euglycemic clamp, isotope dilution technology and indirect calorimetry.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men, with and without a positive family history of schizophrenia.
* 20 kg/m2 < BMI < 26 kg/m2
* Age 20-40 years
* Fasting plasma glucose < 6 mmo/L

Exclusion Criteria:

* FPG > 6 mmol/L
* BMI > 26 kg/m2
* Psychiatric disorders and/or use of antipsychotic or antidepressants drugs at present or in the past.
* Any significant chronic disease
* Renal, hepatic or endocrine disease
* Use of medication known to influence lipolysis and/or glucose metabolism
* Total cholesterol > 7mmol/L and/or triglycerides > 2 mmol/L
* Recent weight changes or attempts to loose weight (> 3 kg weight gain or loss, within the last 3 months)
* Difficulties to insert an intravenous catheter
* Smoking (current)
* Severe claustrophobia (ventilated hood)
* Recent blood donation (within the last 2 months)
* Recent participation in other research projects (within the last 3 months), participation in 2 or more projects in one year
* Extensive sporting activities (more than 10 hours of exercise per week)

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2004-05; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
To determine the effect of subchronic olanzapine and haloperidol treatment on HGO, whole body peripheral glucose disposal, fatty acid flux and fuel oxidation. | 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Hanno Pijl, Phd MD, Study Chair — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands